CLINICAL TRIAL: NCT03708640
Title: A Prospective Randomized Pilot Study to Evaluate the Effect of a Mobile Health Physical Activity Intervention for HIV-associated Frailty
Brief Title: mHealth Physical Activity Trial for Older HIV-infected Adults (mFIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00169068; K23AI108357 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: HIV
Keywords: Frailty; Physical Activity; HIV; Aging; Exercise; mHealth; smartphone; activity tracker; pedometer; text messaging; Short Message Service (SMS)
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Counseling (Placebo Comparator): Group receives baseline physical activity counseling.
  Group does not receive personalized, health coaching via "smart" text messages.
  Interventions: Other: Physical Activity Counseling
- Digital Activity Tracker/Smart Text Messaging (Experimental): Group receives baseline physical activity counseling.
  Group receives personalized, health coaching via "smart" text messages informed by digital activity tracker.
  Interventions: Other: Digital Activity Tracker; Other: Smart Text Messaging; Other: Physical Activity Counseling

INTERVENTIONS:
Other: Digital Activity Tracker — Group wears physical activity tracker and receives physical activity feedback information informed by the tracker
  Arms: Digital Activity Tracker/Smart Text Messaging
Other: Smart Text Messaging — Group receives personalized, health coaching via "smart" text messages
  Arms: Digital Activity Tracker/Smart Text Messaging
Other: Physical Activity Counseling — Group receives baseline counseling on physical activity

SUMMARY:
This pilot study will examine the effect of a mobile health text messaging platform linked to a digital physical activity tracker on physical activity among persons living with HIV and frailty.

DETAILED DESCRIPTION:
HIV is associated with frailty, an important aging-related phenotype associated with adverse clinical outcomes. The investigators propose that personalized health coaching using a digital activity tracker with mobile health text messaging can increase physical activity in this population. The total duration of the intervention will be 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive adults of any gender
* Age 50 years and older
* Frailty score of 2 or greater (at least 1 criteria is slow gait speed or decreased grip strength)
* Ability to provide informed consent

Exclusion Criteria:

* Any physical condition that would prevent or prohibit moderate physical activity
* >3 days per week of moderate or vigorous leisure time activity lasting >30 min/day

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change in Mean daily step count | Baseline, 12 weeks
  Mean daily step count will be assessed using a digital physical activity tracker

SECONDARY OUTCOMES:
Change in Frailty as assessed by the Fried-based physical frailty phenotype | Baseline, 12 weeks
  Frailty evaluated based on the standard 5 point Fried-based frailty phenotype construct (slow gait, weakness, weight loss, exhaustion, low physical activity)
Change in Physical Fitness as assessed by 12 minute walk | Baseline, 12 weeks
  Physical fitness of participants will be assessed by the ability to do a 12 minute walk
Change in Muscle strength as assessed by isokinetic resistance | Baseline, 12 weeks
  Muscle strength evaluated using isokinetic resistance testing on a Biodex system measuring peak torque expressed as foot pounds (lbs)
Percent change in fat mass | Baseline, 12 weeks
  Fat mass will be measured using the dual-energy x-ray absorptiometry (DXA) scan
Percent change in lean mass | Baseline, 12 weeks
  Lean mass will be measured using the dual-energy x-ray absorptiometry (DXA) scan
Change in Physical performance as assessed by the physical performance battery | Baseline, 12 weeks
  Physical performance evaluated with the short physical performance battery
Change in Quality of Life as assessed by the Medical Outcomes Study HIV Health Survey (MOS-HIV) | Baseline, 12 weeks
  The Medical Outcomes Study HIV Health Survey (MOS-HIV) is a brief, comprehensive measure of health-related quality of life. The 35-item questionnaire includes 10 dimensions (pain, physical, role, health perceptions, social and cognitive functioning, energy, mental health, health distress and quality of life). Each dimension is scored on a 0-100 scale (a higher score indicates better health related quality of life). An overall score is obtained through a summation of z scores from each domain.
Change in Interleukin-6 (IL-6) concentration | Baseline, 12 weeks
  Interleukin-6 concentration in pg/ml will be measured at baseline and be compared to the concentration at 12 weeks to assess any change
Change in soluble Tumor Necrosis Factor Receptor 1 (sTNFR1) | Baseline, 12 weeks
  sTNFR1 concentration in ng/ml will be measured at baseline and be compared to the concentration at 12 weeks to assess any change

CONTACTS AND LOCATIONS:
Overall Officials: Damani Piggott, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156